CLINICAL TRIAL: NCT02824653
Title: Allogenic Bone Marrow Mesenchymal Stem Cells Infusion in Patients With Steroid-refractory GVHD- A Phase I/II Clinical Trial
Brief Title: Allogenic Bone Marrow Mesenchymal Stem Cells Infusion in Patients With Steroid-refractory GVHD
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Institute of Blood and Marrow Transplant (NIBMT), Pakistan (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AFBMTC-GVHD-2015
Record Dates: First submitted 2016-06-28; First posted 2016-07-07 (Estimated); Last update posted 2017-01-25 (Estimated); Status verified 2017-01

CONDITIONS: Graft Versus Host Disease
Keywords: acute GVHD; chronic GVHD; steroid-refractory; Mesenchymal Stem Cells
MeSH Terms: conditions — Graft vs Host Disease; Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Mesenchymal Stem Cells (Experimental): The experimental arm is comprised of GVHD patients receiving allogenic bone marrow mesenchymal stem cells
  Interventions: Biological: Mesenchymal Stem Cells

INTERVENTIONS:
Biological: Mesenchymal Stem Cells — Allogenic Human Bone Marrow Mesenchymal Stem Cells (ex-vivo expanded in pooled human platelet lysate)
  Other Names: Allogenic Bone Marrow MSCs

SUMMARY:
Graft versus host disease is a serious and often life-threatening complication in allogeneic haematopoietic stem cell transplantation. Although corticosteroids are the first-choice of treatment in these patients, but about 30-50% patients do not respond to it and develop steroid-refractory GVHD. Mesenchymal stem cells (MSC) have emerged as a promising treatment option in these patients. This phase-I/II clinical trial aims at establishing the safety and clinical efficacy of allogenic ex-vivo cultured MSCs to treat steroid-refractory GVHD in a Pakistani HSCT cohort.

DETAILED DESCRIPTION:
Allogeneic haematopoietic stem cell transplant has become first choice of treatment for many malignant and non malignant haematological disorders. Although great progress has been made to prevent and minimize transplant-associated complications, yet graft versus host disease (GVHD) remains a significant complication affecting these the outcome in these patients. It is a severe inflammatory condition that arises when recipient tissues are attacked by immune mediated donor T cells during transplantation. Acute GVHD predominately affects the skin, upper and lower GI tract, liver and occasionally the eye and oral mucosa, whereas chronic GVHD resembles more with autoimmune disorders in its clinical symptoms. These symptoms can be organ-specific or generalized throughout body.

The pathophysiology of GVHD shows that it has different phases. In first phase i.e., afferent phase, damage to host tissue occurs. In second phase i.e., Induction and expansion phase, donor T cells are triggered and activated by recipient and donor APC as well as the inflammatory cytokines. Activated T cells produce IL-2 and IFN-γ (or Th1 response). Allogeneic immune response is amplified by IL-2, which activates more T cells and natural killer cell responses, triggering macrophages to release TNF-α and further inflammation damages skin and gut. The third phase i.e., effector phase, is characterized by cytotoxic damage against host cells by activated donor T-cell-mediated through Fas-Fas ligand interaction, perforin-granzyme and TNF-α. The latter has a central role in the pathophysiology, stimulating cytokine production (IL-1, IL-6, IL-10, IL-12 and TNF-α). This dysregulation leads to the clinical manifestations of acute GVHD.

The cells involved in GVHD pathophysiology include CD4+ T cells; for maintaining the expansion of CD8+ T cells that mediate GVHD, APCs; these have role in the initiation phase of acute GVHD as described in murine models and Natural killer (NK) cells; contribute to tissue damage in the effector phase by releasing inflammatory cytokines and nitric oxide. However, natural killer cells mediate cell death by two important pathways: Fas-Fas-ligand-mediated apoptosis and perforin-granzyme-B-mediated cytolysis.

HLA differences between donor and recipient are the major predictor of GVHD. Other affecting factors include age, gender mismatch between donor and recipient, minor histocomapatability antigen expression difference(mHA) in otherwise identical HSCT, donor age, source and dose of stem cells (PBSCT greater risk than BM), intensity of conditioning and GVHD prophylaxis.

Steroids are the first line therapy for acute GVHD patients and are standard treatment for grade II-IV acute GVHD. Adverse effects of glucocorticoids include hypertension hyperglycemia and psychosis, immunosuppression, infections, myopathy, osteoporosis and avascular necrosis of bone, cataracts and fat re-distribution etc. If acute GVHD is not improved after 5-7 days treatment with steroids then it is considered as steroid-refractory. Various agents that are being investigated from last two decades as second line therapy include low-dose MTX, MMF, extracorporeal photopheresis, IL-2R targeting, antibody therapy against CD3, CD7, CD25, CD52, CD147, IL-2R, IL-1, and TNF-α (i.e., basiliximab, daclizumab, denileukin, diftitox and alemtuzumab), horse ATG, etanercept, infliximab, and sirolimus and recently infusions of mesenchymal stem cells.

Mesenchymal stem cells (MSCs) are defined as self-renewing, multipotent progenitor cells with potential to differentiate into other cell types of mesodermal origin, such as adipocytes, osteocytes, and chondrocytes. Mesenchymal and Tissue Stem Cell Committee of the International Society for Cellular Therapy developed the minimal criteria for definition of MSCs which is as follows: first, adherence to plastic; Second, positivity for the cell-surface molecules CD105, CD73, and CD90 and negativity for CD45, CD34, CD14 or CD11b, CD79a or CD19, and human leukocyte antigen (HLA)-DR; and third, the ability to differentiate into osteoblasts, adipocytes, and chondroblasts under standard in vitro differentiation conditions. Since Le Blanc and colleagues first reported successful treatment of a patient with severe acute GVHD using third-party haploidentical MSCs in 2004, many clinical trials worldwide have described the benefits of MSC therapy in GVHD.

The proposed project is a phase I/II clinical trial of single group, open label, interventional study design. The objective is to observe the safety and efficacy of intravenous injection of ex-vivo expanded bone marrow mesenchymal cells from a third party donor for treating refractory GVHD. The study will also document the type and frequency of any adverse event or side effects, if discovered.

ELIGIBILITY:
Inclusion Criteria:

* Must fill Informed consent.
* Patient who has undergone allogeneic HSCT and has steroid-refractory grade II-IV acute GVHD.
* Patients who did not respond to treatment options including methylprednisolone, and or cyclosporine A or ATG.
* Patients who despite above mentioned treatment have unresponsive GVHD after 5 days or progressive acute GVHD for more than 72 hours.
* Patients who have received any other treatment and had discontinued for non-responsiveness.

Exclusion Criteria:

* Poor performance status, not expected to survive 5 days.
* Patients with hypersensitivity to penicillin and/or gentamycin.
* Poor compliance.

Ages: 1 Year to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-01; Primary Completion 2016-07 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Incidence of treatment-emergent adverse events and complications [Safety and Tolerability] | 4 weeks
  Safety will be evaluated by reporting any incidence of adverse event, complication and toxicity related to administration of MSCs within 4 weeks of last infusion .
Acute GVHD-restaging [Efficacy] | 4 weeks
  Efficacy of ex-vivo expanded allogenic mesenchymal stem cell infusion will be determined by organ-specific re-staging and global grading of Acute GVHD as per consensus group criteria. Response will be measured as complete response (CR), partial response (PR), stable disease(SD) and progressive disease(PD). CR:acute GVHD symptoms and signs disappear; PR:aGVHD symptoms and signs improve; SD:aGVHD symptoms and signs remain (without improvement or deterioration);PD: aGVHD symptoms and signs deteriorate.
Chronic GVHD-restaging [Efficacy] | 3 months
  Organ-specific scoring and global scoring of chronic GVHD will be done as per NIH consensus criteria of 2014. Treatment response will be measured as complete response (CR), partial response (PR), stable disease(SD) and progressive disease(PD). CR:chronic GVHD symptoms and signs disappear; PR:cGVHD symptoms and signs improve; SD:cGVHD symptoms and signs remain (without improvement or deterioration);PD: cGVHD symptoms and signs deteriorate.

SECONDARY OUTCOMES:
Survival analysis at six months after MSC infusion | 6 months
  Documenting patients' survival status after 6 months of receiving MSC infusion
  To document relapse of hematological malignancies post-MSC infusion.
  Evaluation of late infectious complications or toxicities after MSC infusion.
Incidence free survival at six months after MSC infusion | 6 months
  To document rate of GVHD recurrence in patients after MSC infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Parvez Ahmed, FCPS, MCPS, Principal Investigator — Armed Forces Bone Marrow Transplant Centre, Rawalpindi, Pakistan
Locations (1):
- Armed Forces Bone Marrow Transplant Centre, Rawalpindi, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided